CLINICAL TRIAL: NCT06749626
Title: Progressive Relaxation Exercises Applied After Laparoscopic Cholecystectomy Surgery; Pain Intensity, Physiological Parameters, Anxiety and Its Effect on Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Buse Dinçer, Nurse, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BartınU- SBF- BD- 01
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy Surgery
Keywords: pain; anxiety; physiological parameters; laparoscopic cholecystectomy; progressive relaxation exercise; discharge
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group undergoing progressive relaxation exercise after laparoscopic cholecystectomy surgery (Experimental): Progressive relaxation exercises lasting approximately 30 minutes were applied to the patients in the experimental group, accompanied by the researcher, at the 6th hour, when the nonsteroidal anti-inflammatory drug administered by the clinic was half-done, and at the 10th hour after the surgery.
  Interventions: Other: progressive relaxation exercise
- Group without progressive relaxation exercise after laparoscopic cholecystectomy surgery (No Intervention): Patients in the control group were treated only according to the clinical analgesia protocol.

INTERVENTIONS:
Other: progressive relaxation exercise — Relaxation exercises CD developed by the Turkish Psychologists Association; It consists of muscle exercises, rhythmic breathing and music recital. The CD content, which includes relaxation exercises accompanied by music, was prepared by Psychologist Elif Kabak and voiced by Tülay Bursa. The CD, which includes deep breathing and muscle relaxation exercises, consists of three parts. The first section includes the definition of deep relaxation, the purpose of relaxation exercises and the rules to be considered in exercise practice. In the second part; There are relaxation exercises with audio instructions accompanied by streaming sounds. The third part contains relaxation music without instructions. After the information in the first part of the CD is explained to the patients in the experimental group, the second part, which lasts only approximately 30 minutes, will be administered under the supervision of the researcher. However, since the patients have undergone abdominal surgery, the
  Arms: Group undergoing progressive relaxation exercise after laparoscopic cholecystectomy surgery

SUMMARY:
INTRODUCTION: Among gastrointestinal system diseases, gallbladder diseases are the most common. As is the case after every surgical intervention, changes occur in the patient's homeostasis after laparoscopic cholecystectomy surgery. Studies have shown that more than half of the patients experience moderate to severe pain in the postoperative period. In addition, postoperative pain negatively affects the patients' quality of life by reducing their comfort levels. Progressive relaxation exercises, one of the cognitive-behavioral techniques, aim to gradually contract and relax the patients' muscles. Progressive relaxation exercises; It provides stabilization in physiological parameters by reducing pain caused by muscle tension and increased sympathetic activity after surgery.

At the end of this initiative, it is anticipated that the patient's comfort and satisfaction will increase, the healing process will accelerate, the duration of hospital stay will decrease and, accordingly, hospital care costs will decrease.

PURPOSE: The aim of the thesis study is to determine the progressive relaxation exercises applied after laparoscopic cholecystectomy surgery; To evaluate pain intensity, physiological parameters, anxiety and its effect on discharge.

METHOD: Planned as a randomized controlled experimental study, patients who underwent laparoscopic cholecystectomy surgery at Bartın State Hospital General Surgery Clinic were evaluated according to the algorithm created by the computer program (https://www.randomizer.org/) using numbers from 1 to 102. It will be randomly divided into 2 blocks. A two-block randomization will be made, the first block will be determined as the control group and the second block will be determined as the experimental group. There will be 104 patients in total, 52 in each group. In addition to routine treatment, patients in the experimental group will receive progressive relaxation exercises at the 6th and 10th hour after surgery. After the application, the effect of changes on the patients' pain, physiological parameters, anxiety and discharge will be recorded. 'Data Collection Form', 'Visual Comparison Scale (VAS)', 'Physiological Parameters Monitoring Form', 'State-Trait Anxiety Scale' and 'Readiness for Discharge Scale' will be used to collect data. The analysis of the collected data will be evaluated using the SPSS for Windows 22 program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* No visual or auditory problems,
* Able to speak and understand Turkish,
* No diagnosed psychiatric problems,
* No complications such as bleeding, nausea or vomiting after laparoscopic cholecystectomy surgery,
* Not using patient-controlled analgesia and opioids for postoperative pain control,
* Patients with a pain score ≥4 according to the Visual Comparison Scale will be included.

Exclusion Criteria:

* Those who do not volunteer to participate in the research,
* Having visual or auditory problems,
* Those who cannot speak or understand Turkish,
* Having a diagnosed psychiatric problem,
* Complications such as bleeding, nausea and vomiting occur after laparoscopic cholecystectomy surgery,
* Using patient-controlled analgesia and opioids for postoperative pain control,
* Patients with a pain score <4 according to the Visual Comparison Scale will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale- VAS | For the experimental group, before the progressive relaxation exercise and after the progressive relaxation exercise applied at the 6th and 10th hours, for the control group, before the 6th hour without the progressive relaxation exercise, at the 6th and
  The scale consists of a vertical or horizontal 10 cm straight line and the starting point is 0 and the ending point is 10 cm. The patient is asked to mark where the severity of his pain corresponds to on this line. On the scale, "0" defines the absence of pain and "10" defines the highest unbearable pain.
State-Trait Anxiety Scale | For the experimental group, before the progressive relaxation exercise and after the progressive relaxation exercise applied at the 6th and 10th hours, for the control group, before the 6th hour without the progressive relaxation exercise, at the 6th and
  State Anxiety Scale is a rating scale consisting of 20 items that aims to determine how individuals feel at a certain moment and under conditions. This scale consists of 4-point Likert type answer options; (1) "not at all", (2) "somewhat", (3) "a lot", (4) "completely". After the surgery, the patient is asked to evaluate how he feels "right now" and score the severity of the anxiety states mentioned in each item according to Likert-type expressions. Trait Anxiety Scale is an assessment scale consisting of 20 items that aims to determine how you feel regardless of your current situation. It asks participants to indicate how often they feel anxiety in their general life. The individual is asked to evaluate how he/she "usually" feels by using the following statements on a 4-point Likert-type scale: (1) "almost never", (2) "sometimes", (3) "a lot of the time", (4) "almost always". asked to choose one
Discharge Readiness Scale | It will be applied to patients in both groups the day after surgery.
  The scale has a total of eight items and four subscales. The first and second questions measure how the patient feels during the day, the third and fourth questions measure his knowledge about discharge, the fifth and sixth questions measure how and to what extent he can continue his daily life at home after discharge, and the seventh and eighth questions measure the support he can receive at home after he is discharged. The average total score obtained from the scale is considered very ready for discharge between 9-10, very ready for discharge between 8-8.9, moderately ready between 7-7.9, and low ready if below 7.
Physiological Parameters Monitoring Form | For the experimental group, before the progressive relaxation exercise and after the progressive relaxation exercise applied at the 6th and 10th hours, for the control group, before the 6th hour without the progressive relaxation exercise, at the 6th and
  In the form, patients' systolic and diastolic blood pressure, body temperature, pulse rate, respiratory rate and oxygen saturation are evaluated.
Data Collection Form | The Data Collection Form will be filled out at least 1 hour before the surgery.
  It was prepared in line with the literature information scanned by the researcher and consists of two parts. In the first part, it is about evaluating the sociodemographic characteristics of the patient; It includes age, education level, height-weight, marital status, profession, working status, chronic diseases, constantly used medications and smoking. In the second part, it is about evaluating the clinical characteristics of the patient; It includes questions evaluating the presence of previous surgery, the duration of the surgery, the presence and type of analgesia administered after the surgery, and the date of hospitalization and discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartin State Hospital, Bartın, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want IPD to be shared.